CLINICAL TRIAL: NCT06254521
Title: Neoadjuvant Treatment of Locally Advanced MSS Rectal Cancer With Tislelizumab Combined With CAPOX Regimen: a Prospective, Single-arm, Single-center, Exploratory Phase II Clinical Study
Brief Title: The Effects of Neoadjuvant Tislelizumab Combined With Chemotherapy in Locally Advanced MSS Rectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Hui Li, Deputy chief physician, First Affiliated Hospital of Guangxi Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOYT
Record Dates: First submitted 2024-01-01; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Rectal Cancer; Rectal Cancer Stage II; Rectal Cancer Stage III
Keywords: locally advanced rectal cancer; neoadjuvant; PD-1
MeSH Terms: conditions — Rectal Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Intervention Model Description: Patients with locally advanced rectal cancer who met the inclusion criteria received two or four cycles of Tislelizumab combined Capecitabine and Oxaliplatin regimen chemotherapy and were evaluated by enhanced CT and MRI\TRUS. Then, these patients will receive curative surgery for rectal cancer.
  Interventions:
  Drug: Oxaliplatin Drug: Capecitabine Drug: Tislelizumab Procedure: curative surgery for rectal cancer
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- neoadjuvant Tislelizumab combined with chemotherapy (Experimental): Patients with locally advanced rectal cancer who met the inclusion criteria received two or four cycles of Tislelizumab combined Capecitabine and Oxaliplatin regimen chemotherapy and were evaluated by enhanced CT and MRI\TRUS. Then, these patients will receive curative surgery for rectal cancer.
  Interventions:
  Drug: Oxaliplatin Drug: Capecitabine Drug: Tislelizumab Procedure: curative surgery for rectal cancer
  Interventions: Drug: Tislelizumab combined with chemotherapy

INTERVENTIONS:
Drug: Tislelizumab combined with chemotherapy — Drug: Oxaliplatin Oxaliplatin 130mg/m2 for chemotherapy on Day 1 every 3 weeks and repeat for 2 or 4 cycles. The dose reduction protocol for oxaliplatin-induced toxicity was implemented according to the report in BJC (2018) 118:1322-1328.
  Drug: Capecitabine Oral Capecitabine 1000 mg/m2 twice daily combined with oxaliplatin chemotherapy from Day 1 to Day 14 every 3 weeks and repeat for 2 or 4 cycles. The dose reduction protocol for capecitabine-induced toxicity was implemented according to the report in BJC (2018) 118:1322-1328.
  Drug: Anti-PD-1 Monoclonal Antibody 200 mg on Day 1 every 3 weeks and repeat for 2 or 4 cycles. The incidence of adverse events with Anti-PD-1 Monoclonal Antibodies is relatively low. The PD-1 monoclonal antibody (Tislelizumab) dose adjustment was implemented according to the prescribing information.
  Other Names:
  Tislelizumab
  Procedure: Colectomy The specific surgical approach, whether it be laparoscopic

SUMMARY:
This study aims to elucidate the effects of neoadjuvant Tislelizumab combined with chemotherapy in locally advanced MSS rectal cancer.

DETAILED DESCRIPTION:
The standard treatment for locally advanced rectal cancer is neoadjuvant chemoradiotherapy followed by total mesorectal excision (TME). Pelvic chemoradiotherapy for locally advanced rectal cancer reduces the risk of disease recurrence in the pelvis to less than 10% and has been standard care in North America since 1990.However, it is associated with short-term and long-term toxic effects that can adversely affect quality of life and physical function.

Immunogenic cell death will be enhanced by oxaliplatin-induced immunogenicity and combined with anti-programmed cell death 1 (PD-1) monoclonal antibodies for neoadjuvant therapy. The study will conduct 2 or 4 cycles of Tislelizumab with Oxaliplatin and Capecitabine, followed by TME surgery. This study's primary endpoint is the proportion of pCR in the pathological specimens of surgically resected tumors.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old and ≤70 years old.
* Pathologically diagnosed MSS ((confirmed by microsatellite stable detection or next-generation target sequencing) or (confirmed by immunohistochemistry)) colon adenocarcinoma.
* The lower edge of the tumor is less than 12cm from the anus as measured by colonoscopy and MRI,or TRUS.
* It was confirmed by magnetic resonance imaging (MRI) or intracavitary ultrasound of the rectum as T3-4 or N+, and M0 by enhanced CT.
* The ECOG physical status score is 0-1.
* Life expectancy is expected to be more than 1 year.
* First diagnosis, no previous anti-tumor treatment received, and no chemotherapy contraindications.
* Appropriate organ function is defined as follows: Hemoglobin level ≥ 90g/L, Neutrophil count ≥ 1.5×10^9/L, Platelet count ≥ 75×10^9/L, Serum total bilirubin ≤ 1.5× the upper limit of normal (UNL), Aspartate aminotransferase (AST) ≤ 2× UNL, Alanine aminotransferase (ALT) ≤ 3× UNL, Serum creatinine ≤ 1.5× UNL.
* Informed consent, able to understand the study protocol and willing to participate in the study, and will provide written informed consent.

Exclusion Criteria:

* Early rectal cancer (T1-2N0M0); The lower margin of the tumor was less than 5cm from the anus and T4. APR(combined abdominal perineal resection) is required;
* Multifocal colorectal cancer.
* Tumor obstruction or high risk of obstruction, bleeding, and/or perforation requiring emergency surgery or stent placement.
* Cannot tolerate chemotherapy or immunotherapy, such as but not limited to bone marrow suppression.
* History of malignant tumors, except for basal cell carcinoma, papillary thyroid carcinoma, and various in situ cancers.
* Acute exacerbation of important organ diseases (such as but not limited to COPD, coronary heart disease, and renal insufficiency) and/or severe acute infectious diseases (such as but not limited to hepatitis, pneumonia, and myocarditis), ASA score > 3 points.
* Mental disorders, illiteracy, or language communication barriers that prevent the understanding of the study protocol.
* Peripheral sensory neuropathy, unable to receive oxaliplatin-based chemotherapy.
* Continuous use of glucocorticoids for more than 3 days within 1 month prior to signing the informed consent form, or having comorbidities requiring the use of glucocorticoid therapy.
* Unable to undergo enhanced CT examination
* Pregnancy or lactation.
* Refused to participate in this study.
* Other situations in which the researcher deems unsuitable for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-22 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate | 7days of postoperative pathological examination
  the proportion of tumor regression grades 0 (TRG0, disappearance of tumor cells) in the pathological specimens of surgically resected tumors

SECONDARY OUTCOMES:
Complete Clinical Response(cCR) rate | 5 days before surgery
  cCR:After non-surgical antitumor therapy, physical examination and auxiliary examination(CT and MRI ) found no local evidence of tumor residue.
3-year disease-free survival(DFS) rate | 36 months from date of the patient signs the informed consent form
  DFS:From date of the patient signs the informed consent form until the date of earliest occurrence of the patient's tumor recurrence or death, whichever came first.assessed up to 36 months.CT, MRI and colonoscopy were used to evaluate tumor recurrence.
3-year overall survival(OS) rate | 36 months from date of the patient signs the informed consent form
  OS:From the date of the patient signs the informed consent form until the date of the patient's death.assessed up to 36 months.
the rate of adverse events(AEs) | From the first day of immunotherapy until 6 months after the end of treatment
  Adverse events (NCI CTC AE 5.0) that occurred from the first day of chemotherapy to one day of treatment end (up to half a year).
the rate of immune-related adverse events(irAEs) | From the first day of immunotherapy until 6 months after the end of treatment
  Immune-related adverse events (NCCN irAEs (2021)) that occurred from the first day of immunotherapy to one day of treatment end (up to half a year).
the rate of R0 resection | 7 days of postoperative pathological examination
  the rate of a microscopically margin-negative resection, in which no gross or microscopic tumor remains in the primary tumor bed
the rate of surgical complication during or after operation | From the day of surgery to 30 days after the operation
  From the day of surgery to 30 days after the operation, including intraoperative and postoperative complications(bleeding，anastomotic fistula，intestinal obstruction，Anastomotic stenosis，Surgical site infection（SSI），urinary retention，sexual dysfunction)
Retain anal proportions | immediately after the surgery
  The proportion of cases with anal retention in all patients undergoing surgery
3-year local recurrence rate | 36 months from date of the patient signs the informed consent form
  From the date of the patient signs the informed consent form until the date of the local recurrence, assessed up to 36 months. CT, MRI and colonoscopy were used to evaluate local recurrence.

OTHER OUTCOMES:
T lymphocyte | 1-7 days before treatment, 1-7 days before surgery, 1 day after surgery, 3 months after surgery, and 6 months after surgery
  Cells with cellular immune function. The types and counts of T cells are analyzed using flow cytometry
Molecular pathological analysis of tumor tissue | Tumor tissue was obtained 1 month before treatment and analyzed 36 months after treatment
  Whole exome gene sequencing is performed on tumor specimens to analyze the gene status

CONTACTS AND LOCATIONS:
Overall Officials: Hui Li, Professor, Study Chair — First Affiliated Hospital of Guangxi Medical University
Locations (1):
- The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: Yes
We will share the research proposal after registration; Primary study endpoint data were shared 15 days after surgery; All data will be shared 3 years after enrollment
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: We will share the research proposal after registration; Primary study endpoint data were shared 15 days after surgery; All data will be shared 3 years after enrollment
Access Criteria: Clinician or researcher
URL: https://clinicaltrials.gov/